CLINICAL TRIAL: NCT04805645
Title: Clinical Characteristics & Risk Factors for Mortality of COVID-19 Patients Admitted Into Intensive Care Unit in Hospital Queen Elizabeth
Brief Title: Risk Factors for Mortality for COVID-19 Admitted to an Intensive Care Unit
Acronym: ICUCOVID-KK
Status: Terminated | Type: Observational
Why Stopped: Study was unable to begin due to clinicians too busy with handling COVID-19 cases
Sponsor: Clinical Research Centre, Malaysia (Other)
Collaborators: Hospital Queen Elizabeth, Malaysia (Other Government)
Responsible Party: Sponsor
Other Study IDs: ICUCOVID-KK
Record Dates: First submitted 2021-03-16; First posted 2021-03-18 (Actual); Last update posted 2023-09-01 (Actual); Status verified 2023-08

CONDITIONS: Covid19; Critically Ill
Keywords: COVID-19; Critically ill; Mortality Day 28
MeSH Terms: conditions — COVID-19; Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Non-Survivors: Participants who had Critically-ill COVID-19 and admitted to the Intensive Care Unit which died before or on day 28 post ICU admission
  Interventions: Other: No intervention (Retrospective Cohort Observational)
- Survivors: Participants who had Critically-ill COVID-19 and admitted to the Intensive Care Unit whom are still alive on day 28 post ICU admission

INTERVENTIONS:
Other: No intervention (Retrospective Cohort Observational) — No intervention as this study is a Retrospective Cohort Observational
  Groups: Non-Survivors

SUMMARY:
Studying clinical characterization of critically ill COVID-19 patients in a single center Studying Risk factors for Day 28 Mortality in COVID-19 patients admitted to intensive care unit

DETAILED DESCRIPTION:
An observational study looking into clinical characterization of the novel Coronavirus Disease 2019 (COVID-19) in patients admitted, critically ill, into Intensive Care Unit of Hospital Queen Elizabeth between 1st October 2020 until 31st January 2021. Analysis also would be looking into the risk factors into Day 28 mortality of these patients

ELIGIBILITY:
Inclusion Criteria:

* All patients admitted to the ICU in Hospital Queen Elizabeth, Kota Kinabalu between 1st October 2020 until 31st January 2021
* Confirmed COVID-19 Positive using RT-PCR or RTK-Ag either before or during admission in ICU

Exclusion Criteria:

* Patients that were admitted in ICU suspected to have COVID-19 and died in ICU which subsequently to be COVID-19 negative

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: All patients admitted to the ICU in Hospital Queen Elizabeth, Kota Kinabalu between 1st October 2020 until 31st January 2021, which confirmed to have via PCR testing or Rapid Test Antigen are positive for PCR
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2021-04-01 (Actual); Study Completion 2021-05-01 (Actual)

PRIMARY OUTCOMES:
Mortality | 28 days
  Died before or on Day 28 after ICU admission

SECONDARY OUTCOMES:
Oxygen supplementation requirement | day 28
  Requirement of oxygen supplementation on day 28 after icu admission

CONTACTS AND LOCATIONS:
Overall Officials: Kean Khang Fong, Principal Investigator — Hospital Queen Elizabeth, Malaysia
Locations (1):
- Hospital Queen Elizabeth, Kota Kinabalu, Malaysia

IPD SHARING:
Plan to Share IPD: No